CLINICAL TRIAL: NCT05798416
Title: Effect of Supplement of CO2 Using Novel Portable Device on Exercise Performance at High Altitude
Brief Title: Effect of Inhalation of Low Dose CO2 on Exercise Performance at High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yuan-Ming Luo, Professor, State Key Laboratory of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020 No.37
Record Dates: First submitted 2023-03-10; First posted 2023-04-04 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: High Altitude; Inhalation; Gas; Acute Mountain Sickness
Keywords: High altitude; Exercise performance; CO2 inhalation
MeSH Terms: conditions — Altitude Sickness; Respiratory Aspiration; Mucopolysaccharidosis IV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise under inhalation of CO2 (Active Comparator): Subjects will perform shuttle walk test under inhalation of low concentration of CO2 supplied by a novel device at high altitude.
  Interventions: Drug: Exercise under inhalation CO2
- Exercise under inhalation of ambient air (Placebo Comparator): Subjects will perform shuttle walk test under inhalation of ambient air at high altitude.
  Interventions: Other: Exercise under inhalation ambient air

INTERVENTIONS:
Drug: Exercise under inhalation CO2 — Participants perform shuttle walk test at high altitude while using the novel portable device for inhalation of CO2
  Other Names: inhalation of low dose CO2
  Arms: Exercise under inhalation of CO2
Other: Exercise under inhalation ambient air — Participants perform shuttle walk test at high altitude while inhaling ambient air
  Arms: Exercise under inhalation of ambient air

SUMMARY:
High altitude (>2400 m) is associated with decreased atmosphere pressure leading to hypoxia which in turn impairs exercise capacity and causes acute mountain sickness (AMS). It is noted that adding CO2 might be beneficial to improve hypoxia and exercise performance at high altitude. However, no device is currently available that can supply a constant low dose of CO2 during free movement at high altitude. We have recently invented a portable device which is small and light enough for supplement of low dose CO2 during field exercise at high altitude.

DETAILED DESCRIPTION:
Objective: To determine whether the supplement of low-dose CO2 by the novel device could improve exercise performance at high altitude.

Methods: The lowlanders (<500m) who have no history of travelling to high altitude (>1000m) a year before the study will be recruited. And the subjects who are high-altitude residents and have not left high altitude over the last twelve months will also be recruited for the study. Subjects will be randomly and blindly given either CO2 mixed with air or air alone during endurance shuttle walking test (ESWT). Blood gases will be measured before and after inhalation of CO2. ESWT time, ventilation per minute (VE), blood oxygen saturation (SPO2), and end-tidal CO2 concentration (ETCO2) will be measured during exercise and will be compared during inhalation of CO2 and during inhalation of ambient air.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy lowlanders (<500m) who have no history to travel to high altitude (>1000m) a year before the study.
2. Healthy high altitude (4500m) residents who have not left the inhabited area over the last twelve months before the study.

Exclusion Criteria:

1. Subjects with cardiovascular diseases, respiratory diseases and neuromuscular diseases which could affect exercise.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Change of the distance in walking test | 48 hours
  Changes in walking distance under inhalation of CO2 and ambient air

CONTACTS AND LOCATIONS:
Overall Officials: Yuanming Luo, PhD, Principal Investigator — The Affiliated Hospital og Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after the paper of this study publishing.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be shared after the paper of this study publishing.
Access Criteria: After the paper of this study publishing